CLINICAL TRIAL: NCT05487911
Title: Cortical rTMS as a Treatment for Depression
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Hyuntaek Oh, PhD, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-51886
Record Dates: First submitted 2022-06-27; First posted 2022-08-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: MDD subjects enrolled will receive TMS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- rTMS (Experimental): 20 sessions of rTMS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — 4 weeks of active rTMS (total of up to 20 sessions)

SUMMARY:
Major depressive disorder (MDD) is a leading cause of disability worldwide with a 19% lifetime prevalence in the United States. Dysfunctional reward processing (e.g., the loss of pleasure) is one of the core features of MDD. Common treatments of MDD include psychological therapies (e.g., cognitive behavioral therapy), medication (e.g., bupropion, sertraline), and psychological therapies and medication combined, but they may not address the function of the reward circuit in MDD. These treatments often do not improve depressive symptoms in MDD patients who are classified as having treatment-resistant depression, and they may be unlikely to respond to further medication trials. Transcranial magnetic stimulation (TMS) is a non-invasive brain stimulation that enables us to selectively excite or inhibit neural activity. Multiple TMS pulses given consecutively are known as repetitive TMS (rTMS), and the primary clinical location for applying rTMS is the left dorsolateral prefrontal cortex (dlPFC) for treatment of MDD. Many of these studies have shown that rTMS to the dlPFC may result in decreased depressive symptoms, but is only partially effective (response and remission rates of 41.2 and 35.3%, respectively). This evidence supports the importance of evaluating the efficacy of rTMS in other brain regions, such as the orbitofrontal cortex (OFC), in the treatment of MDD rather than in the dlPFC.

DETAILED DESCRIPTION:
The OFC is functionally connected to other cortical brain regions (e.g., prefrontal and parietal cortices) but also to subcortical areas in the dorsal striatum, a core reward circuitry region. The OFC is structurally connected to the medial forebrain bundle (MFB), deep brain stimulation (DBS) target for MDD, and the OFC may in fact be the mediator of anti-depressant effect. The functional connectivity between the OFC and those subcortical brain regions also plays an important role in addiction and suicide behaviors, which are MDD's most common comorbidities. Thus, it is clear that investigators need a better understanding of the therapeutic mechanisms using non-invasive brain stimulation (e.g., TMS) treatment to the OFC as applied to MDD patients. As such, the investigators propose to use a combination of interleaved TMS-fMRI, a novel method to observe and characterize causal manipulations of functional neural circuits, targeting the OFC and resting state fMRI to longitudinally study depressive symptoms and depression-related symptoms (e.g., addiction, suicidal behaviors) changes in MDD patients.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female aged 18-60 years old
* Meets MDD criteria
* Has depressive symptoms according to the Patients Health Questionnaire (PHQ)-9 or Hamilton Depression Rating Scale (HDRS) or Snaith-Hamilton Pleasure Scale (SHAPS)
* Be able to verbalize understanding of consent form, able to provide written informed consent, and verbalize willingness to complete study procedures
* Female subjects must be non-nursing and not pregnant at the times of fMRI experiments and TMS treatment
* Has no contraindications to MRI (pacemaker, cochlear implants, metal in eyes, other metal implants, etc.); Meets the pre- screening MRI questions provided by the Center for Advanced MR Imaging (CAMRI)
* Has no contraindications to TMS (any types of non-removable metal in their head except the mouth, or within 12 inches of the coil, etc.); Meets the pre-screening TMS safety questionnaire (Transcranial Magnetic Stimulation Adult Safety Screen - TASS)

Exclusion Criteria:

* In the opinion of the clinician and/or the research team, be expected to fail to complete the study protocol due to not tolerable to receive TMS
* Unable to understand the design and requirements of the study
* Unable to sign informed consent for any reason
* Has an unstable medical condition, including AIDS, acute hepatitis, active TB, unstable cardiac disease, unstable diabetes, hepatic or renal insufficiency
* Female subjects who are pregnant or nursing
* Contraindications to MRI (pacemaker, cochlear implants, metal in the eye, other metal implants, etc.): Do not meet the pre-screening MRI questions provided by the CAMRI at BCM
* Contraindications to TMS (any types of non-removable metal in their head except the mouth, or within 12 inches of the coil, etc.): Do not meet the pre-screening TMS safety questionnaire (TASS). Additional exclusion criteria for the TMS experiments are based on the recommendations described by the international consensus panel on brain stimulation.
* Non-English speaking subjects (we do not have the staff and/or resources to include other language).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-04 (Estimated); Study Completion 2027-08-04 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity of orbital frontal cortex (OFC) | 20 days
  Functional connectivity of OFC changes after receiving TMS treatment
Outcome Changes in MDD subjects | 20 days
  The relationship between the functional connectivity changes and clinical outcome changes in MDD

CONTACTS AND LOCATIONS:
Locations (1):
- The Menninger Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Bromet EJ. The epidemiology of depression across cultures. Annu Rev Public Health. 2013;34:119-38. doi: 10.1146/annurev-publhealth-031912-114409. PMID 23514317
- [Background] Admon R, Pizzagalli DA. Dysfunctional Reward Processing in Depression. Curr Opin Psychol. 2015 Aug 1;4:114-118. doi: 10.1016/j.copsyc.2014.12.011. PMID 26258159
- [Background] Forbes EE, Christopher May J, Siegle GJ, Ladouceur CD, Ryan ND, Carter CS, Birmaher B, Axelson DA, Dahl RE. Reward-related decision-making in pediatric major depressive disorder: an fMRI study. J Child Psychol Psychiatry. 2006 Oct;47(10):1031-40. doi: 10.1111/j.1469-7610.2006.01673.x. PMID 17073982
- [Background] Nutt DJ. Care of depressed patients with anxiety symptoms. J Clin Psychiatry. 1999;60 Suppl 17:23-7; discussion 46-8. PMID 10446738
- [Background] Horst WD, Preskorn SH. Mechanisms of action and clinical characteristics of three atypical antidepressants: venlafaxine, nefazodone, bupropion. J Affect Disord. 1998 Dec;51(3):237-54. doi: 10.1016/s0165-0327(98)00222-5. PMID 10333980
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Stewart JW, Nierenberg AA, Thase ME, Ritz L, Biggs MM, Warden D, Luther JF, Shores-Wilson K, Niederehe G, Fava M; STAR*D Study Team. Bupropion-SR, sertraline, or venlafaxine-XR after failure of SSRIs for depression. N Engl J Med. 2006 Mar 23;354(12):1231-42. doi: 10.1056/NEJMoa052963. PMID 16554525
- [Background] Hallett M. Transcranial magnetic stimulation: a primer. Neuron. 2007 Jul 19;55(2):187-99. doi: 10.1016/j.neuron.2007.06.026. PMID 17640522